CLINICAL TRIAL: NCT04771403
Title: A Randomized, Two-way, Cross-over Study to Assess the Efficacy of an MPC Exercise-enabled Closed-loop System vs FMPD Exercise-enabled Closed-loop System
Brief Title: Two Way Crossover Closed Loop Study MPC vs FMPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Jessica Castle, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19973
Record Dates: First submitted 2021-01-27; First posted 2021-02-25 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes
Keywords: glucose sensor; automated insulin delivery systems
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- FMPD AP system (Experimental): Participants will use the FMPD AP system for automated insulin delivery for a 76 hour study visit.
  Interventions: Device: FMPD AP algorithm
- MPC AP System (Experimental): Participants will use the MPC AP system for automated insulin delivery for a 76 hour study visit.
  Interventions: Device: MPC AP system
- Dexcom G6 Training Arm (Experimental): Participants will use the Dexcom G6 CGM system within the MPC AP system to generate sensor glucose data during a 7 day period.
  Interventions: Device: Dexcom G6 Continuous Glucose Monitoring (CGM) System

INTERVENTIONS:
Device: FMPD AP algorithm — The Fading Memory Proportional Derivative (FMPD) insulin infusion algorithm determines insulin delivery rates based on proportional error, defined as the difference between the current CGM level and the target CGM level, and the derivative error, defined as the rate of change of the CGM. The FMPD algorithm utilizes derivative and proportional glucose errors to determine delivery rates of insulin.
  Arms: FMPD AP system
Device: MPC AP system — The Model Predictive Control (MPC) insulin infusion algorithm contains a model within the controller that takes as an input the aerobic metabolic expenditure in addition to the CGM and meal inputs. The algorithm uses heart rate and accelerometer data collected on the patient's body to calculate metabolic expenditure. The metabolic expenditure then acts on the model for the insulin dynamics, whereby more energy expenditure and longer duration exercise can lead to a more substantial effect of insulin on the CGM.
  Arms: MPC AP System
Device: Dexcom G6 Continuous Glucose Monitoring (CGM) System — The Dexcom G6 CGM measures interstitial glucose through a sensor transmitter. This glucose value is reported to the MPC algorithm during this intervention.
  Arms: Dexcom G6 Training Arm

SUMMARY:
An artificial pancreas (AP) is a control system for automatic insulin delivery. Our group has implemented a fading memory proportional derivative controller (FMPD) for use within an AP control system which has been evaluated in clinical studies. However, the long action of insulin (90 minutes for peak action) makes it challenging to control insulin with a classical proportional derivative system. The study described within this protocol is designed to test the effectiveness of a new model-predictive control (MPC) AP that modulates insulin delivery based on estimated activity level. The potential benefit of this type of AP is that it handles exercise not as a discrete event, but it automatically adjusts insulin delivery based on estimated activity level calculated at every 5 minute cycle. This type of algorithm may significantly improve glucose control over our FMPD AP, which is designed only to detect exercise when activity level goes above a threshold for a specific duration of 45 minutes.

DETAILED DESCRIPTION:
Participants will undergo two approximately 76 hour studies. During each of these intervention visits, participants will wear an Omnipod to deliver insulin and a Dexcom G6 CGM to measure glucose. The CGM system will provide sensed glucose data every 5 minutes. Sensed glucose data will be wirelessly transmitted via Bluetooth Low Energy (BTLE) from the Dexcom G6 transmitter to the Samsung master controller every five minutes. The smart phone will wirelessly communicate via BTLE to an Omnipod through an Omnipod PDM. During one of the studies, glucose will be controlled using the MPC AP. During another study, glucose will be controlled using the FMPD AP. The AP system will receive activity data through a Polar M600 watch worn by the participant.

Participants will arrive at the clinic at approximately 7am for the inpatient visits. Participants will eat breakfast, lunch and dinner in the clinic. Participants will perform activities of daily living and exercise using an aerobic exercise video. Participants will discharge at 7pm to go home for the remainder of the study visit and perform one exercise video session at home. Participants will return to OHSU on Day 4 for removal of all devices. The exception to this is for the first 8 participants using the MPC AP. These participants will stay at the research clinic during the day and go home to sleep each night (7pm-7am).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female participants 21 to 50 years of age.
* Physically willing and able to perform aerobic exercise (as determined by the investigator after reviewing the participant's activity level)
* Current use of an insulin pump for at least 3 months with stable insulin pump settings for >2 weeks.
* Lives with another person age 18 or older who will be present while participant exercises at home and that can attend the training on using the system.
* Lives within 40 miles of OHSU main campus.
* HbA1c ≤ 10% at screening.
* Total daily insulin requirement is less than 139 units/day.
* Current use of a phone or other device so can be contacted by study staff off-campus
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as reported by the OHSU laboratory).
* Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
* Hematocrit of less than 36% for men, less than 32% for women.
* Hypertensive participants with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg despite treatment or who have treatment-refractory hypertension (e.g. requiring four or more medications).
* History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. Participants will complete a hypoglycemia awareness questionnaire. Participants will be excluded for four or more R responses.
* History of diabetes ketoacidosis during the prior 6 months prior to screening visit, as diagnosed on hospital admission or as judged by the investigator.
* Adrenal insufficiency.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to aspart or lispro insulin.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Beta blockers or non-dihydropyridine calcium channel blockers.
* Current use of any medication intended to lower glucose other than insulin (ex. use of liraglutide).
* A positive response to any of the questions from the Physical Activity Readiness Questionnaire with one exception: participant will not be excluded if he/she takes a single blood pressure medication that doesn't impact heart rate and blood pressure is controlled on the medication (blood pressure is less than 140/90 mmHg).
* Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort.
* Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the participant's safety or compliance with the protocol.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jacobs, PhD, Principal Investigator — Oregon Health and Science University; Jessica Castle, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobs PG, Resalat N, Hilts W, Young GM, Leitschuh J, Pinsonault J, El Youssef J, Branigan D, Gabo V, Eom J, Ramsey K, Dodier R, Mosquera-Lopez C, Wilson LM, Castle JR. Integrating metabolic expenditure information from wearable fitness sensors into an AI-augmented automated insulin delivery system: a randomised clinical trial. Lancet Digit Health. 2023 Sep;5(9):e607-e617. doi: 10.1016/S2589-7500(23)00112-7. Epub 2023 Aug 3. PMID 37543512

RESULTS

PARTICIPANT FLOW:
Groups:
- MPC to FMPD: The randomization order for participants in this arm was Model Predictive Control (MPC) followed by Fading-Memory Proportional Derivative (FMPD). Each visit was about 76 hours and included an inpatient and outpatient portion. The first 8 participants using the MPC remained as inpatients in clinic during the day and went home with system turned off at night (7pm-7am).
- FMPD to MPC: The randomization order for participants in this arm was Fading-Memory Proportional Derivative (FMPD) followed by Model Predictive Control (MPC). Each visit was about 76 hours and included an inpatient and outpatient portion. The first 8 participants using the MPC remained as inpatients in clinic during the day and went home with system turned off at night (7pm-7am).
Period: Dexcom Training Visit (1 Week)
Arm/Group | MPC to FMPD | FMPD to MPC
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: First Rest Period (1-12 Weeks)
Arm/Group | MPC to FMPD | FMPD to MPC
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: First Intervention (~76 Hours)
Arm/Group | MPC to FMPD | FMPD to MPC
Started | 13 | 12
Completed | 9 | 10
Not Completed | 4 | 2
Not completed — FMPD study stopped after 7 hours: Pod occlusion with hyperglycemia (data not analyzed) | 0 | 1
Not completed — MPC study stopped after 8 hours due to algorithm safety concerns (data not analyzed) | 1 | 0
Not completed — MPC Study stopped after 34 hrs for safety due to high ketones (data analyzed) | 1 | 0
Not completed — MPC study stopped after 61 hrs due to cloud server issues (data analyzed) | 1 | 0
Not completed — MPC study stopped after 32 hours due to algorithm safety concerns (data analyzed) | 1 | 0
Not completed — FMPD study stopped after 6 hours due to algorithm safety concerns (data not analyzed) | 0 | 1
Period: Second Rest Period (1-10 Weeks)
Arm/Group | MPC to FMPD | FMPD to MPC
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Subject withdrawn before completing FMPD study due to safety concerns due to keto diet | 1 | 0
Period: Second Intervention Visit (~76 Hours)
Arm/Group | MPC to FMPD | FMPD to MPC
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — FMPD study stopped after 25 hrs due to stopping rules for hypoglycemia (data analyzed) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MPC to FMPD: The randomization order for participants in this arm was Model Predictive Control (MPC) followed by Fading-Memory Proportional Derivative (FMPD). Each visit was about 72 hours and included a 12 hour inpatient and 60 hour outpatient portion.
- FMPD to MPC: The randomization order for participants in this arm was Fading-Memory Proportional Derivative (FMPD) followed by Model Predictive Control (MPC). Each visit was about 72 hours and included a 12 hour inpatient and 60 hour outpatient portion.
- Total: Total of all reporting groups
Arm/Group | MPC to FMPD | FMPD to MPC | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (8.9) | 33.4 (8.9) | 34.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 9 | 22
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time With Sensed Glucose <70 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 70 mg/dl using Dexcom sensor across the duration of the 12 hour inpatient stay (either Day 3 or Day 1 MPC vs. Day 1 FMPD).
Time Frame: 12 hour inpatient stay (either Day 3 or Day 1 MPC vs. Day 1 FMPD)
Population: Out of 25 participants enrolled, the MPC study cancelled after 8 hours was not analyzed, the other three MPC studies that were cancelled after 30+ hours were analyzed. Two FMPD studies were cancelled the first day, 6 or 7 hours in and one FMPD study never happened as participant was withdrawn, so three FMPD studies were not analyzed. The other FMPD study that was cancelled after 28 hours was analyzed.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage of time | 2.5 (7.0) | 1.3 (2.9)

2. Secondary Outcome: Percent of Time With Sensed Glucose Between 70-180 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values between 70-180 mg/dl using Dexcom sensor across both arms.
Time Frame: During each 76 hour intervention study (2 total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage of time | 75.5 (10.7) | 71.2 (16.1)

3. Secondary Outcome: Percent of Time With Sensed Glucose Between 70 - 180 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values between 70-180 mg/dl using Dexcom sensor across the duration of the 12 hour inpatient stay (either Day 3 or Day 1 MPC vs. Day 1 FMPD).
Time Frame: 12 hour inpatient stay (either Day 3 or Day 1 MPC vs. Day 1 FMPD)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage of time | 59.4 (23.1) | 63.2 (23.9)

4. Secondary Outcome: Percent of Time With Sensed Glucose Between 70 - 180 mg/dl After Exercise
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values between 70-180 mg/dl using Dexcom sensor across both arms from the start of the in-clinic exercise session until the start of the next meal.
Time Frame: start of the in-clinic exercise session until the start of the next meal, approximately 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage of time | 81 (22) | 87 (17)

5. Secondary Outcome: Percent of Time With Sensed Glucose <70 mg/dl After Exercise
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 70 mg/dl using Dexcom sensor across both arms from the start of the in-clinic exercise session until the start of the next meal.
Time Frame: start of the in-clinic exercise session until the start of the next meal, approximately 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage of time | 4.9 (14.4) | 1.4 (4.2)

6. Secondary Outcome: Number of Carbohydrate Treatments
Description: Assess the mean number of carbohydrate treatments (defined as 15 or 20 grams of carbohydrate) across both arms.
Time Frame: During each 76 hour intervention study (2 total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: carbohydrate treatments/day
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
carbohydrate treatments/day | 1.03 (1.34) | 0.65 (0.84)

7. Secondary Outcome: Mean Sensed Glucose
Description: Assess the mean sensed glucose from the Dexcom G6 reported sensor glucose values across both arms. The Dexcom G6 CGM updates every 5 minutes with a new CGM value for 10 days. The Dexcom G6 reads values between 40-400 mg/dL with an urgent low alert at 55 mg/dl, a low and high alert when CGM goes above or below the alert thresholds set by the user. Physiologically relevant thresholds for the Dexcom G6 CGM sensor glucose values are less than 55 mg/dl, less than 70 mg/dl, above 180 mg/dl and above 250 mg/dl. The Dexcom G6 target range is 70-180 mg/dl.
Time Frame: During each 76 hour intervention study (2 total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
mmol/L | 8.5 (0.9) | 8.8 (1.3)

8. Secondary Outcome: Coefficient of Variation of Glucose
Description: Assess the coefficient of variation of glucose from the Dexcom G6 reported sensor glucose values across both arms. The Dexcom G6 CGM updates every 5 minutes with a new CGM value for 10 days. The Dexcom G6 reads values between 40-400 mg/dL with an urgent low alert at 55 mg/dl, a low and high alert when CGM goes above or below the alert thresholds set by the user. Physiologically relevant thresholds for the Dexcom G6 CGM sensor glucose values are less than 55 mg/dl, less than 70 mg/dl, above 180 mg/dl and above 250 mg/dl. The Dexcom G6 target range is 70-180 mg/dl.The target coefficient of variation is 33% or lower.
Time Frame: During each 76 hour intervention study (2 total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage | 28.4 (5.9) | 29.6 (6.9)

9. Secondary Outcome: Percent of Time With Sensed Glucose <54 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 54 mg/dl using Dexcom sensor across both arms
Time Frame: During each 76 hour intervention study (2 total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage of time | 0.13 (0.33) | 0.05 (0.15)

10. Secondary Outcome: Percent of Time With Sensed Glucose >180 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values greater than 180 mg/dl using Dexcom sensor across both arms
Time Frame: During each 76 hour intervention study (2 total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
percentage of time | 23.2 (10.9) | 27.8 (16.0)

11. Secondary Outcome: Mean Amount of Insulin Delivered Per Day (in Units/Day)
Description: Assess the mean amount of insulin delivered per day by the Omnipod through the AP system study in units/kg across both arms.
Time Frame: During each 76 hour intervention study (2 total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | FMPD AP System | MPC AP System
Number analyzed (Participants) | 22 | 24
units/day | 40.8 (16.0) | 44.6 (22.6)

ADVERSE EVENTS:
Time Frame: 12 months
Description: All participants that began/started the Dexcom training visit or an MPC or FMPD arm visit are included in the adverse events. The numbers from the participant flow indicate that 25 subjects began the Dexcom training visit, 25 subjects began an MPC visit and 24 subjects began an FMPD visit.
Groups:
- Dexcom G6 Training Arm: Participants will use the Dexcom G6 CGM with the MPC AP algorithm for acquiring sensor glucose values.
Arm/Group | MPC AP System | FMPD AP System | Dexcom G6 Training Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 0/24 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPC AP System (N=25) | FMPD AP System (N=24) | Dexcom G6 Training Arm (N=25)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Back Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
High ketones (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Ketones measured by Precision Xtra blood ketone meter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT04771403/Prot_SAP_000.pdf